CLINICAL TRIAL: NCT04285918
Title: Evaluation of Prevalence and Clinical Impact of Atrial Fibrillation in Elderly Patients With Cryptogenic Stroke and High-Risk Patent Foramen Ovale
Acronym: DefenseElderly
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Jae-Kwan Song, Jae-Kwan Song, Asan Medical Center
Other Study IDs: 2019-1112
Record Dates: First submitted 2020-02-25; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Cryptogenic Stroke; High Risk Patent Foramen Ovale
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Patients ≥60 y/o with ESUS and PFO that is likely to have causative role (high-risk anatomical feature)
  Interventions: Procedure: Percutaneous device closure
- Cohort B: Patients ≥60 y/o with ESUS without PFO, or with non-high risk PFO

INTERVENTIONS:
Procedure: Percutaneous device closure — If there is no relevant AF detected for 6 months during intermittent follow-up or ICM, device closure of PFO is recommended for high-risk PFOs but is decided ultimately at the discretion of the attending physician. If there is any relevant AF identified from ICM or other modalities during follow-up, adequate secondary prevention with anticoagulants should be carried out. All this process and decision making should be a part of routine clinical practice.
  Groups: Cohort A

SUMMARY:
The purpose of DEFENSE-ELDERLY is to identify the prevalence of AF and evaluate the clinical impact of AF in elderly ESUS patients and no other known sources of stroke besides a high-risk patent foramen ovale, and compare it with elderly ESUS patients without high-risk PFO (no PFO or non-high risk PFOs)

DETAILED DESCRIPTION:
The purpose of DEFENSE-ELDERLY is to identify the prevalence of AF and evaluate the clinical impact of AF in elderly ESUS patients and no other known sources of stroke besides a high-risk patent foramen ovale, and compare it with elderly ESUS patients without high-risk PFO (no PFO or non-high risk PFOs)

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥60 y/o with ESUS and PFO that is likely to have causative role (high-risk anatomical feature) (cohort A)
* Patients ≥60 y/o with ESUS without PFO, or with non-high risk PFO (cohort B)
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the institutional review board
* Patients who are scheduled to have implantable cardiac monitoring

Exclusion Criteria:

* Transient ischemic attack
* Lacunar infarction (infarction at subcortical area with a lesion diameter less than 2cm on MR)
* Presence of complex aortic atheroma (≥4mm in plaque thickness or presence of mobile components)
* Presence of ≥50% luminal stenosis (extra- or intracranial) in arteries supplying the ischemic area
* Unwillingness or inability to comply with the procedures described in this protocol
* Life expectancy < 1 years for any non-cardiac or cardiac causes

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥60 y/o with ESUS and PFO that is likely to have causative role (high-risk anatomical feature) (cohort A) and Patients ≥60 y/o with ESUS without PFO, or with non-high risk PFO (cohort B)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-10-02 (Actual); Primary Completion 2024-10-02 (Estimated); Study Completion 2024-10-02 (Estimated)

PRIMARY OUTCOMES:
Paroxysmal AF episodes > 30 seconds detected with intermittent recordings or ≥ 2 minutes during ICM within 6 months | Enrollment to 6 months
  Paroxysmal AF episodes > 30 seconds detected with intermittent recordings or ≥ 2 minutes during ICM within 6 months

SECONDARY OUTCOMES:
Paroxysmal AF episodes > 30 seconds detected with intermittent recordings or ≥ 2 minutes during ICM within 36 months | Enrollment to 36 months
  Paroxysmal AF episodes > 30 seconds detected with intermittent recordings or ≥ 2 minutes during ICM within 36 months
Paroxysmal AF episodes > 30 seconds detected with intermittent recordings or ≥ 6 minutes during ICM at 6 months and 36 months | 6 months to 36 months
  Paroxysmal AF episodes > 30 seconds detected with intermittent recordings or ≥ 6 minutes during ICM at 6 months and 36 months
Rates of percutaneous device closure, prescription of anticoagulants (warfarin or direct oral anticoagulants) | Enrollment to 36 months
  Rates of percutaneous device closure, prescription of anticoagulants (warfarin or direct oral anticoagulants)
Recurrent stroke or TIA | Enrollment to 36 months
  Recurrent stroke or TIA
All-cause death, Vascular Death | Enrollment to 36 months
  All-cause death, Vascular Death

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided